CLINICAL TRIAL: NCT00098995
Title: A Phase I Study Of Tirapazamine In Combination With Radiation And Weekly Cisplatin In Patients With Locally Advanced Cervical Cancer
Brief Title: Tirapazamine, Cisplatin, and Radiation Therapy in Treating Patients With Stage IB, Stage II, Stage III, or Stage IVA Cervical Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: PMCC-2004/354; CDR0000393978 (Registry Identifier: PDQ (Physician Data Query)); NCI-5485
Record Dates: First submitted 2004-12-08; First posted 2004-12-09 (Estimated); Last update posted 2013-06-26 (Estimated); Status verified 2006-11

CONDITIONS: Cervical Cancer
Keywords: stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; cervical adenocarcinoma; cervical adenosquamous cell carcinoma; cervical squamous cell carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Tirapazamine; Brachytherapy; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: tirapazamine
Radiation: brachytherapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as tirapazamine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Tirapazamine may help cisplatin kill more tumor cells by making tumor cells more sensitive to the drug. Radiation therapy uses high-energy x-rays to kill tumor cells. Tirapazamine may also make tumor cells more sensitive to radiation therapy. Giving radiation therapy in different ways together with combination chemotherapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of tirapazamine when given together with cisplatin and radiation therapy in treating patients with stage IB, stage II, stage III, or stage IVA cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose and the recommended phase II and III dose of tirapazamine when combined with cisplatin and radiotherapy in patients with Stage IB-IVA squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma of the cervix.
* Determine the safety and tolerability of this regimen in these patients.

Secondary

* Determine failure-free survival of patients treated with this regimen.
* Determine overall survival of patients treated with this regimen.
* Determine time to locoregional failure in patients treated with this regimen.
* Determine patterns of failure for the site of first failure in patients treated with this regimen.
* Determine the 12-week post-treatment complete response rate in patients treated with this regimen.

OUTLINE: This is a multicenter, dose-escalation study of tirapazamine.

Patients receive tirapazamine IV over 2 hours on day 1 of weeks 1-5 and on days 3 and 5 of weeks 1 and 2 (cohort 2 only), OR days 3 and 5 of weeks 1-4 (cohort 3 only). Patients also receive cisplatin IV over 1 hour on day 1 of weeks 1-6. Patients concurrently undergo external beam radiotherapy once daily on days 1-5 for 5-5.5 weeks. After completion of chemoradiotherapy, patients undergo low-dose brachytherapy (up to 2 implants within an 8-week period) OR high-dose brachytherapy twice weekly for 5 treatments. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of tirapazamine until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. At least 10 patients are treated at the MTD.

Patients are followed at 2, 4, and 8 weeks, at 3 and 6 months, every 3 months for 2 years, and then every 6 months for 2 years.

PROJECTED ACCRUAL: A total of 3-22 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma of the cervix

  * Stage IB, IIA, IIB, III, or IVA disease
* No evidence of involvement of para-aortic nodes by CT scan, MRI, fluorodeoxyglucose positron emission tomography, or lymphadenectomy

  * Involvement of common iliac nodes allowed
* No evidence of distant metastases

PATIENT CHARACTERISTICS:

Age

* Any age

Performance status

* ECOG 0-2

Life expectancy

* More than 6 months

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3

Hepatic

* Bilirubin < 1.25 times upper limit of normal (ULN)
* AST and ALT ≤ 3 times ULN

Renal

* Calculated creatinine clearance ≥ 60 mL/min OR
* Glomerular filtration rate ≥ 60 mL/min

Cardiovascular

* No significant cardiac disease that would preclude IV fluid load required for administration of cisplatin
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other

* No symptomatic peripheral neuropathy ≥ grade 2
* No clinically significant sensori-neural hearing impairment interfering with activities of daily living or requiring a hearing aid

  * Audiometric changes alone of any severity allowed
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to tirapazamine or cisplatin
* No other invasive malignancy within the past 5 years except nonmelanoma skin cancer
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* No other concurrent uncontrolled illness
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent epoetin alfa
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* No concurrent pegfilgrastim

Chemotherapy

* No prior chemotherapy for another malignancy

Endocrine therapy

* Not specified

Radiotherapy

* No prior pelvic or abdominal radiotherapy for another malignancy
* No prior radiotherapy to ≥ 15% of bone marrow-bearing areas
* No concurrent intensity-modulated radiotherapy
* No concurrent interstitial brachytherapy

Surgery

* Not specified

Other

* No prior treatment for invasive cervical cancer
* No other concurrent therapeutic investigational agents
* No other concurrent anticancer therapy
* No concurrent systemic retinoids
* No concurrent amifostine
* No concurrent combination antiretroviral therapy for HIV-positive patients

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2004-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of tirapazamine
Safety and tolerability

SECONDARY OUTCOMES:
Failure-free survival
Overall survival
Patterns of failure for the site of first failure (local-regional, distant, or both)
Complete response rate at 12 weeks following study completion
Hypoxia by 18F-azomycinarabinoside (FAZA) PET scan at baseline and 12 wks following completion of radiotherapy correlated w/ obj. tumor response by PET- fludeoxyglucose F 18 (FDG) and local-regional failure

CONTACTS AND LOCATIONS:
Overall Officials: Danny Rischin, MD, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia
- Princess Margaret Hospital, Toronto, Ontario, Canada